CLINICAL TRIAL: NCT06853730
Title: Regional Distribution Mapping of Lymph Node Metastasis in Epithelial Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Xu Huishan (Other)
Responsible Party: Sponsor-Investigator, Xu Huishan, Research Assistant, Ovarian Cancer Study Group, Sun Yat-sen University, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: SYSU-LNM-OVCA01
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer
Keywords: Lymph Node Metastasis
MeSH Terms: conditions — Ovarian Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-metastasis Group: This group consists of ovarian cancer patients without lymph node metastasis. By comparing with the metastasis group, we aim to identify the clinical factors that differentiate patients with and without metastasis.
- Metastasis Group: This group includes ovarian cancer patients with lymph node metastasis. We will analyze the clinical characteristics and metastasis pathways of these patients to identify clinical factors associated with metastasis.Based on the clinical factors (such as the location of the primary tumor, stage of cancer, etc.), we further subgroup the metastatic patients (e.g., based on the side of the primary tumor). This analysis aims to explore whether there are specific patterns or pathways of lymph node metastasis in these subgroups.

SUMMARY:
The goal of this observational study is to investigate the metastatic pathways of lymph node involvement in ovarian cancer patients. The main question it aims to answer is: • What are the sequential patterns of lymph node metastasis in ovarian cancer, and are there specific clinical factors associated with different metastatic pathways? Participants diagnosed with ovarian cancer who have undergone lymphadenectomy as part of their standard treatment will have their postoperative pathological lymph node involvement analyzed. The study will retrospectively collect and analyze patient data, including lymph node metastasis patterns, to identify potential progression routes.

ELIGIBILITY:
Inclusion Criteria:i) initial diagnosis and tumor cytoreductive surgery performed at the First Affiliated Hospital of Sun Yat-sen University; ii) confirmed postoperative pathology of epithelial ovarian cancer; iii) available lymph node status; and iv) accessible clinical features, including preoperative ultrasound and blood biochemistry tests

Exclusion Criteria: i) initial diagnosis or surgical treatment conducted at other hospitals; ii) absence of imaging results (CT/PET-CT/MRI) or postoperative pathology results for lymph node status. iii) presence of other cancers; and iv) incomplete medical history

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with epithelial ovarian cancer at the First Affiliated Hospital of Sun Yat-sen University from January 2014 to December 2022 were included in this retrospective study. The inclusion criteria were as follows: i) initial diagnosis and tumor cytoreductive surgery performed at the First Affiliated Hospital of Sun Yat-sen University; ii) confirmed postoperative pathology of epithelial ovarian cancer; iii) available lymph node status; and iv) accessible clinical features, including preoperative ultrasound and blood biochemistry tests. The exclusion criteria were: i) initial diagnosis or surgical treatment conducted at other hospitals; ii) absence of imaging results (CT/PET-CT/MRI) or postoperative pathology results for lymph node status. iii) presence of other cancers; and iv) incomplete medical history
Sampling Method: Non-Probability Sample
Enrollment: 654 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of lymph node metastasis in ovarian cancer patients and its association with clinical factors. | From enrollment to 6 months post-surgery
  The primary goal of this study is to determine the frequency of lymph node metastasis in patients with ovarian cancer and identify clinical factors associated with the occurrence of metastasis.

IPD SHARING:
Plan to Share IPD: No